CLINICAL TRIAL: NCT04768881
Title: A Phase 2 Open-Label Multicenter Study to Evaluate the Safety and Efficacy of Selinexor in Combination With Pembrolizumab in Recurrent Advanced Melanoma
Brief Title: Safety and Efficacy of Selinexor in Combination With Pembrolizumab in Recurrent Advanced Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was terminated due to a lack of sufficient anti-melanoma tumor signal for the combination of selinexor + pembrolizumab.
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XPORT-MEL-033
Record Dates: First submitted 2021-02-22; First posted 2021-02-24 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Locally Advanced Unresectable or Metastatic Melanoma
Keywords: Karyopharm; Locally advanced unresectable or metastatic melanoma; KPT-330; Recurrent advanced melanoma; Selinexor; Pembrolizumab
MeSH Terms: conditions — Melanoma | interventions — selinexor; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Primary resistance to Initial CPI Therapy (Experimental): Participants will receive a dose of 80 milligrams (mg) selinexor orally once weekly (QW) and a dose of pembrolizumab 400 mg intravenously (IV) once in every six weeks (Q6W), both on Day 1 of a 6-week cycle until progressive disease (PD), intolerable toxicity or withdrawal from the study, whichever occurs first.
  Interventions: Drug: Selinexor; Drug: Pembrolizumab
- Arm B: Acquired Resistance to Initial CPI Therapy (Experimental): Participants will receive a dose of 80 mg selinexor orally once weekly (QW) and a dose of pembrolizumab 400 mg IV Q6W, both on Day 1 of a 6-week cycle until PD, intolerable toxicity or withdrawal from the study, whichever occurs first.
  Interventions: Drug: Selinexor; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Selinexor — Dose and formulation: 80 mg (4 tablets of 20 mg)
  Other Names: KPT-330; XPOVIO®
Drug: Pembrolizumab — Dose and formulation: 400 mg (25 milligrams per milliliter [mg/mL]) Solution
  Other Names: KEYTRUDA®

SUMMARY:
Approximately 40 participants with locally advanced or metastatic melanoma will be enrolled in 20 sites in the United States into 1 of the following 2 arms: Primary resistance to initial checkpoint inhibitor (CPI) therapy in Arm A and Acquired resistance to initial CPI therapy in Arm B. Participants who have disease progression (PD) after discontinuation of CPIs, especially in neoadjuvant or adjuvant therapy, will be considered to have acquired resistance in this study. Participants will receive study treatment (Selinexor and Pembrolizumab) until PD, intolerable toxicity or withdrawal from the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to (≥) 18 years at the time of informed consent.
* Participant must have a histologically confirmed diagnosis of locally advanced unresectable stage III or metastatic stage IV melanoma not amenable to local therapy.

  1. Participants must have confirmed PD per Response Evaluation Criteria in Solid Tumors (RECIST) on or within 12 weeks of the last dose of anti-PD-1/L1 monotherapy or combination therapy (including relatlimab or other anti-LAG-3 mAb) per Society for Immunotherapy in Cancer Guidelines (Kluger,2020).
  2. Arm A (primary resistance): participant has disease progression after receiving at least 6 weeks of prior anti-PD-1/L1 mAb with the best response as PD, or stable disease (SD) less than (<) 6 month (participants with a partial response [PR] or complete response [CR] who have disease progression within 6 months will be considered to have primary resistance in this study).
  3. Arm B (secondary/acquired resistance): participant has disease progression after receiving at least 6 months of prior anti-PD-1/L1 mAb with the best response as CR, PR, or SD greater than (>) 6 months (participants who have disease progression after neoadjuvant or adjuvant therapy, will be considered to have secondary resistance in this study).
  4. Participants who progress on or within 12 weeks after elective discontinuation of anti-PD-1/L1 mono or combination treatment in the absence of PD or treatment limiting toxicity must have confirmed PD per RECIST.
* Participants should have at least 1 prior line of CPI therapy but no more than 2.
* Measurable disease according to RECIST v1.1.
* Participants with stable previously treated brain metastases are permitted in this study.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to (≤) 1.
* Adequate bone marrow function at screening, defined as:

  1. Absolute neutrophil count (ANC) ≥1.5 * 10^9 per liter (L).
  2. Hemoglobin ≥10 gram per deciliter (gm/dL) (≥6.2 millimoles per liter [mmol/L]).
  3. Platelet count ≥100 * 10^9/L.
* Serum direct bilirubin ≤1.5 * upper limit of normal (ULN); aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 * ULN (with confirmed liver metastases: AST and ALT ≤5 * ULN).
* Calculated creatinine clearance (CrCl) ≥15 milliliters per minute (mL/min) based on the Cockcroft and Gault formula.
* Female participants of childbearing potential must have a negative serum pregnancy test at screening and agree to use highly effective methods of contraception throughout the study and for at least four months following the last dose of study treatment. Childbearing potential excludes: Age >50 years and naturally amenorrhoeic for >1 year, or previous bilateral salpingo-oophorectomy, or hysterectomy.
* Male participants who are sexually active must use highly effective methods of contraception throughout the study and for at least four months following the last dose of study treatment. Male participants must agree not to donate sperm during the study treatment period.
* Written informed consent signed in accordance with federal, local, and institutional guidelines.

Exclusion Criteria:

* Metastatic uveal or ocular melanoma.
* Active central nervous system (CNS) metastases or other CNS (e.g., meningeal) involvement.
* Participants must have resolution or improvement of immune-mediated treatment related adverse reactions related to prior treatment(s) to Grade ≤1 without steroid maintenance therapy or his or her previous baseline prior to the corresponding CPI therapy

  a. History of immune-mediated treatment related adverse reactions leading to discontinuation of prior anti-programmed death protein 1 (PD-1), anti-programmed death protein ligand 1 (PD-L1), or anti programmed death protein ligand 2 (PD-L2) monoclonal antibodies (mAbs) or severe hypersensitivity reaction to any mAb or any excipients which in the opinion of the Investigator precludes future use of anti-PD-1/PDL1 therapy.
* Concurrent systemic steroid therapy higher than physiologic dose (>10 milligrams per day [mg/day] of prednisone or equivalent).
* Previous treatment with selinexor or other exportin 1 (XPO1) inhibitors.
* Insufficient time since or not recovered from procedures or anti-cancer therapy, defined as:

  1. Not recovered from major surgery ≤28 days prior to Day 1 dosing. Minor procedures, such as biopsies, dental work, or placement of a port or intravenous (IV) line for infusion are permitted.
  2. Have ongoing clinically significant anti-cancer therapy-related toxicities Common Terminology Criteria for Adverse Events (CTCAE) Grade >1. In specific cases, participants whose toxicity has stabilized or with Grade 2 non-hematologic toxicities can be allowed following documented approval by the Sponsor's Medical Monitor
  3. Had last dose of previous anti-cancer therapy ≤14 days prior to Day 1 dosing
  4. Palliative radiotherapy >14 days prior to the study is allowed
  5. Received investigational drugs in other clinical trials within 28 days, or 5 half-lives of the investigational drug (whichever is shorter), prior to Cycle 1 Day 1 (C1D1).
* Live-attenuated vaccine (e.g., nasal spray influenza vaccine) ≤14 days prior to the intended C1D1.
* Impairment of gastrointestinal (GI) function or GI disease that could significantly alter the absorption of selinexor (e.g., vomiting, or diarrhea that is CTCAE version 5.0 grade >1).
* Life expectancy less than (<) 4 months based on the opinion of the Investigator
* Active pneumonitis requiring steroid therapy.
* Uncontrolled (i.e., clinically unstable) infection requiring parenteral antibiotics, antivirals, or antifungals within 7 days prior to first dose of study treatment; however, prophylactic use of these agents is acceptable (including parenteral).
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the participant's safety, prevent the participant from giving informed consent, or being compliant with the study procedures.
* Female participants who are pregnant or lactating.
* Active hepatitis B virus treated with antiviral therapy for hepatitis B within 8 weeks with a viral load >100 international units per milliliter (IU/mL).
* Untreated hepatitis C virus positive without documentation of negative viral load per institutional standard.
* Human immunodeficiency virus positive with CD4+T-cells ≤350 cells per microliter, positive viral load per institutional standard, and a history of acquired immunodeficiency syndrome defining opportunist infections in the last year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - UCLA, Los Angeles, California
  - TOI Clinical Research, Pasadena, California
  - BRCR Global, Plantation, Florida
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Great Plains Health, North Platte, Nebraska
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York Oncology Hematology, Albany, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - OH Care Clinical Trials, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Texas Oncology-Austin Central, Austin, Texas
  - Texas Oncology - Baylor Sammons Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 13 sites in United States of America from 12 May 2021 to 22 September 2023.
Pre-assignment Details: A total of 15 participants were enrolled and received the study treatment. The study was stopped prematurely due to a lack of sufficient anti-tumor signal for the selinexor/pembrolizumab combination treatment in participants with advanced or metastatic melanoma.
Groups:
- Arm A: Primary Resistance to Initial Checkpoint Inhibitor (CPI) Therapy: Participants with advanced or metastatic melanoma were primary resistance to initial CPI therapy received a dose of 80 milligrams (mg) (4 tablets of 20 mg) selinexor orally once weekly (QW) and a dose of pembrolizumab 400 mg intravenously (IV) once in every six weeks (Q6W), both on Day 1 of a 6-week cycle (each cycle = 42 days) until progressive disease (PD), intolerable toxicity or withdrawal from the study, whichever occurred first.
- Arm B: Acquired Resistance to Initial CPI Therapy: Participants with advanced or metastatic melanoma had acquired resistance to initial CPI therapy received a dose of 80 mg (4 tablets of 20 mg) selinexor orally QW and a dose of pembrolizumab 400 mg IV Q6W, both on Day 1 of a 6-week cycle (each cycle = 42 days) until PD, intolerable toxicity or withdrawal from the study, whichever occurred first.
Period: Overall Study
Arm/Group | Arm A: Primary Resistance to Initial Checkpoint Inhibitor (CPI) Therapy | Arm B: Acquired Resistance to Initial CPI Therapy
Started | 9 | 6
Completed | 0 | 0
Not Completed | 9 | 6
Not completed — Completed Study Follow-up | 0 | 2
Not completed — Death | 3 | 2
Not completed — Study Terminated by Sponsor | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population consisted of all participants who received at least one dose of any study treatment.
Groups:
- Arm A: Primary Resistance to Initial CPI Therapy: Participants with advanced or metastatic melanoma where primary resistance to initial CPI therapy received a dose of 80 mg (4 tablets of 20 mg) selinexor orally QW and a dose of pembrolizumab 400 mg IV Q6W, both on Day 1 of a 6-week cycle (each cycle = 42 days) until PD, intolerable toxicity or withdrawal from the study, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Arm A: Primary Resistance to Initial CPI Therapy | Arm B: Acquired Resistance to Initial CPI Therapy | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (13.95) | 53.7 (12.40) | 58.3 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 6 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Assessed as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: ORR was defined as the percentage of participants who achieved complete response (CR) or partial response (PR). ORR was assessed by RECIST 1.1 as defined by the Investigator based on radiologic criteria. Per RECIST 1.1 criteria, CR was defined as disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to less than (<)10 millimeter (mm). PR was defined as at least a 30 percentage (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of randomization until the documentation of CR or PR, whichever occurs first (up to 24 months)
Population: mITT population consisted of all participants who received at least one dose of any study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Primary Resistance to Initial CPI Therapy | Arm B: Acquired Resistance to Initial CPI Therapy
Number analyzed (Participants) | 9 | 6
Percentage of participants | 33.3 [7.5 to 70.1] | 16.7 [0.4 to 64.1]

2. Secondary Outcome: Progression-free Survival (PFS) as Per RECIST v 1.1
Description: PFS was defined as time from date of first treatment to the date of first confirmed progressive disease (PD), assessed by RECIST 1.1 is objectively documented or death due to any cause. As per RECIST 1.1 criteria, PD was defined as at least a 20% increase in the sum of the longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: From the date of randomization until disease progression or death, due to any cause (up to 24 months)
Population: mITT population consisted of all participants who received at least one dose of any study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Primary Resistance to Initial CPI Therapy | Arm B: Acquired Resistance to Initial CPI Therapy
Number analyzed (Participants) | 9 | 6
Months | 3.75 [2.14 to NA] — Upper range of 95% CI could not be estimated due to higher number (>50%) of censored participants. | 6.24 [2.10 to NA] — Upper range of 95% CI could not be estimated due to higher number (>50%) of censored participants.

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of first study treatment until death due to any cause. If death event did not occur during the follow-up period, the participant was censored at the date of discontinuation from the study (i.e. withdrawal of consent), or date of last participating visit (e.g., a telephone contact with participant status being alive) on or before database cutoff date, whichever occurs first.
Time Frame: From the date of first study treatment up to death (up to 24 months)
Population: mITT population consisted of all participants who received at least one dose of any study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Primary Resistance to Initial CPI Therapy | Arm B: Acquired Resistance to Initial CPI Therapy
Number analyzed (Participants) | 9 | 6
Months | NA [8.31 to NA] — Median and upper range of 95% CI could not be estimated due to insufficient number of participants with event | NA [13.08 to NA] — Median and upper range of 95% CI could not be estimated due to insufficient number of participants with event

4. Secondary Outcome: Complete Response Rate (CRR)
Description: Complete response rate was defined as percentage of participants who had achieved a complete response (CR) per RECIST 1.1. As per RECIST version 1.1, CR was defined as disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduced in the short axis to <10 mm.
Time Frame: Up to 101 weeks
Population: mITT population consisted of all participants who received at least one dose of any study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Primary Resistance to Initial CPI Therapy | Arm B: Acquired Resistance to Initial CPI Therapy
Number analyzed (Participants) | 9 | 6
Percentage of participants | 22.2 [2.8 to 60.0] | 16.7 [0.4 to 64.1]

5. Secondary Outcome: Duration of Response (DOR) as Per RECIST v 1.1
Description: DOR was defined as the time from first occurrence of CR or PR until the first date of PD per RECIST version 1.1 or death. Per RECIST 1.1 criteria, CR was defined as disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD was defined as at least a 20% increase in the sum of the longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: From first occurrence of CR or PR until disease progression or death, whichever occurs first (up to 24 months)
Population: mITT population consisted of all participants who received at least one dose of any study treatment. Only those participants who had confirmed response were included in the analysis. Here, "overall number of participants analyzed" signifies those who had response to DOR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Primary Resistance to Initial CPI Therapy | Arm B: Acquired Resistance to Initial CPI Therapy
Number analyzed (Participants) | 3 | 1
Months | NA [1.61 to NA] — Median and upper range of 95% CI could not be estimated due to higher number (>50%) of censored participants. | NA [NA to NA] — Median and 95% CI could not be estimated due to higher number (100%) of censored participants.

6. Secondary Outcome: Percentage of Participants With Disease Control Rate (DCR) as Per RECIST v 1.1
Description: Disease control rate was defined as percentage of participants who have a response of CR, PR, or at least 12 continuous weeks of stable disease (SD) as per RECIST v 1.1. As per RECIST v 1.1 before PD or initiating a new antineoplastic therapy, CR was defined as disappearance of all target lesions; any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (at least a 20% increase in the sum of diameters of target lesions) taking as reference the smallest sum diameters while on study. Percentage values were rounded off.
Time Frame: Up to 24 months
Population: mITT population consisted of all participants who received at least one dose of any study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Primary Resistance to Initial CPI Therapy | Arm B: Acquired Resistance to Initial CPI Therapy
Number analyzed (Participants) | 9 | 6
Percentage of participants | 44.4 [13.7 to 78.8] | 50.0 [11.8 to 88.2]

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. A TEAE was defined as those AEs that develop or worsen after the first dose of study drug. TEAEs included both serious and non-serious TEAEs.
Time Frame: From start of the study treatment up to 24 months
Population: Safety population consisted of all enrolled participants who had received at least one dose of both study treatments.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Primary Resistance to Initial CPI Therapy | Arm B: Acquired Resistance to Initial CPI Therapy
Number analyzed (Participants) | 9 | 6
Participants
  Participants with TEAEs | 9 | 6
  Participants with Serious TEAEs | 3 | 2

8. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Parameters
Description: Clinical laboratory parameters included clinical chemistry, hematology and urinalysis. Number of participants with clinically significant laboratory abnormalities which were deemed clinically significant by the investigator were reported.
Time Frame: From start of the study treatment up to 24 months
Population: Safety population consisted of all enrolled participants who had received at least one dose of both study treatments.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Primary Resistance to Initial CPI Therapy | Arm B: Acquired Resistance to Initial CPI Therapy
Number analyzed (Participants) | 9 | 6
Participants
  Clinical Chemistry | 0 | 0
  Hematology | 0 | 0
  Urinalysis | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs included body temperature, blood pressure (systolic blood pressure and diastolic blood pressure). Measurements were made after the participant had been resting supine for a minimum of 5 minutes. The clinically significant change assessment was based on investigator's judgment. Number of participants with clinically significant change from baseline in vital signs values were reported.
Time Frame: From start of the study treatment up to 24 months
Population: Safety population consisted of all enrolled participants who had received at least one dose of both study treatments.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Primary Resistance to Initial CPI Therapy | Arm B: Acquired Resistance to Initial CPI Therapy
Number analyzed (Participants) | 9 | 6
Participants
  Systolic Blood Pressure | 0 | 0
  Diastolic Blood Pressure | 0 | 0
  Body Temperature | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Changes in Physical Examination
Description: Number of participants with clinically significant physical examination abnormalities including general appearance, dermatological, head, eyes, ears, nose, throat, respiratory, cardiovascular, abdominal, lymph nodes, musculoskeletal, and neurological examinations. Number of participants with clinically significant physical examination abnormalities which were deemed clinically significant by the investigator were reported.
Time Frame: From start of the study treatment up to 24 months
Population: Safety population consisted of all enrolled participants who had received at least one dose of both study treatments.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Primary Resistance to Initial CPI Therapy | Arm B: Acquired Resistance to Initial CPI Therapy
Number analyzed (Participants) | 9 | 6
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Severity of Adverse Events Assessed Using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Description: AEs are graded using the following criteria using Common Terminology Criteria for Adverse events v5.0: Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL; Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL; Grade 4: Life-threatening consequences; urgent intervention indicated; Grade 5: Death related to AE.
Time Frame: From start of the study treatment up to 24 months
Population: Safety population consisted of all enrolled participants who had received at least one dose of both study treatments.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Primary Resistance to Initial CPI Therapy | Arm B: Acquired Resistance to Initial CPI Therapy
Number analyzed (Participants) | 9 | 6
Participants
  Grade 1 | 0 | 0
  Grade 2 | 5 | 2
  Grade 3 | 4 | 4
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of the study treatment up to 24 months
Description: Safety population consisted of all enrolled participants who had received at least one dose of both study treatments.
Arm/Group | Arm A: Primary Resistance to Initial CPI Therapy | Arm B: Acquired Resistance to Initial CPI Therapy
All-Cause Mortality (participants affected / at risk) | 3/9 | 2/6
Serious Adverse Events (participants affected / at risk) | 3/9 | 2/6
Other Adverse Events (participants affected / at risk) | 9/9 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Primary Resistance to Initial CPI Therapy (N=9) | Arm B: Acquired Resistance to Initial CPI Therapy (N=6)
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Primary Resistance to Initial CPI Therapy (N=9) | Arm B: Acquired Resistance to Initial CPI Therapy (N=6)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 2
Anaemia (Blood and lymphatic system disorders) | 4 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 2
Dacryostenosis acquired (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 6
Constipation (Gastrointestinal disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 5 | 1
Oedema peripheral (General disorders) | 2 | 1
Asthenia (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Ear infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0
Weight decreased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0
Carbon dioxide decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 2 | 2
Dysgeusia (Nervous system disorders) | 0 | 3
Cognitive disorder (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Mood altered (Psychiatric disorders) | 1 | 0
Panic disorder (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Adnexa uteri cyst (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was stopped prematurely due to a lack of sufficient anti-tumor signal for the selinexor/pembrolizumab combination treatment in participants with advanced or metastatic melanoma.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/81/NCT04768881/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT04768881/SAP_001.pdf